CLINICAL TRIAL: NCT02187380
Title: Studying the Impact of Medication Counselling by Community Pharmacists in Patients Starting a Treatment With Antidepressants
Acronym: SIMCA
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Sophie Liekens, M Psy, KU Leuven
Other Study IDs: B32220109082; s52518 (Registry Identifier: Clinical Trail Center (CTC), UZ Leuven)
Record Dates: First submitted 2014-07-08; First posted 2014-07-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Depression; Antidepressant
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control group: Pharmacists received no depression training, delivered usual care to patients starting a new treatment with depression.
- Intervention group: Pharmacists received a depression training day and provided structured medication counselling to patients starting a new treatment with antidepressants

SUMMARY:
The objective of the SIMCA study was to analyse the impact of structured medication counselling by community pharmacists on medication adherence, economic, clinical and humanistic outcomes of depressed primary care patients who started a new treatment with antidepressants.

A clustered RCT was set up in the Surplus Network, a pharmacy chain in Flanders, Belgium. At the time of the start of the study, the Surplus Network included 97 pharmacies, in all five Flemish provinces, including Brussels. During pre-trial meetings, all pharmacists were informed about the SIMCA-study and instructed how to approach eligible patients.

Randomisation was obtained at the pharmacy level by a computerized random-number generator, following a permuted block design (1:1). The Surplus Network contains a number of local pharmacy chains; stratiﬁcation was used to ensure equal distribution within local pharmacy chains.

Pharmacists in the intervention group were trained in communication skills related to depression treatment counselling in groups of no more than 10 participants over a single day. In total, 10 training days were scheduled between November and December, 2010.

Patients were eligible for inclusion in the study if they started using at least one antidepressant drug, if they were at least 18 years old, if they were able to understand and complete Dutch questionnaires and if they could be reached by telephone for follow-up. "Starting" was defined as not having been prescribed antidepressants over the last six months, which was checked in the pharmacy records. If the patient gave verbal consent to the pharmacist, to be contacted by the research team, the patient was provided with written and oral information about the SIMCA project and a consent form. At the same time an automatic e-mail was generated from the pharmacy software to inform the research team about the patient's willingness to be contacted about the study. The patient was contacted by the research team, as soon as possible to give more information about the study, to ask for informed consent and to schedule a first telephone survey interview. If the patient wished to participate, he/she completed the consent form, and sent it back with the included postage-paid envelope addressed to the research team. Upon receipt of the consent form, the recruited patient's prescribing doctor was contacted and asked to complete and return a brief questionnaire to provide the diagnosis and its severity related to prescribing antidepressants.

Telephone survey interviews based on validated scales were used to collect data at the start of treatment (as close as possible to the time of recruitment), after one month, three months and six months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* able to understand and complete Dutch questionnaires
* could be reached by telephone for follow-up

Exclusion Criteria:

* used antidepressants over the last six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care patients with a new prescription for antidepressants in Flanders, Belgium.
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2010-06; Primary Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Medication adherence | 1 month after start of antidepressants treatment
  Medication adherence measured by the MMAS-8
Medication adherence | 3 months after start of antidepressants treatment
  Medication adherence measured by the MMAS-8
Medication adherence | 6 months after start of antidepressants treatment
  Medication adherence measured by the MMAS-8

SECONDARY OUTCOMES:
Economic outcomes | at the start of antidepressants treatment
  Economic outcomes are measured by the WPAI
Economic outcomes | 1 month after the start of antidepressants treatment
  Economic outcomes are measured by the WPAI
Economic outcomes | 3 months after the start of antidepressants treatment
  Economic outcomes are measured by the WPAI
Economic outcomes | 6 months after the start of antidepressants treatment
  Economic outcomes are measured by the WPAI
Clinical outcomes | at the start of antidepressants treatment
  Clinical outcomes are measured by the HADS
Clinical outcomes | 1 month after the start of antidepressants treatment
  Clinical outcomes are measured by the HADS
Clinical outcomes | 3 months after the start of antidepressants treatment
  Clinical outcomes are measured by the HADS
Clinical outcomes | 6 months after the start of antidepressants treatment
  Clinical outcomes are measured by the HADS
Beliefs about medicines | At the start of antidepressants treatment
  Patients' beliefs about medicines are measured by the BMQ
Beliefs about medicines | 1 month after the start of antidepressants treatment
  Patients' beliefs about medicines are measured by the BMQ
Beliefs about medicines | 3 months after the start of antidepressants treatment
  Patients' beliefs about medicines are measured by the BMQ
Beliefs about medicines | 6 months after the start of antidepressants treatment
  Patients' beliefs about medicines are measured by the BMQ
Satisfaction with the pharmacist | At the start of antidepressants treatment
  Patients' satisfaction with the pharmacist is measured by the SWiP
Satisfaction with the pharmacist | 1 month after the start of antidepressants treatment
  Patients' satisfaction with the pharmacist is measured by the SWiP
Satisfaction with the pharmacist | 3 months after the start of antidepressants treatment
  Patients' satisfaction with the pharmacist is measured by the SWiP
Satisfaction with the pharmacist | 6 months after the start of antidepressants treatment
  Patients' satisfaction with the pharmacist is measured by the SWiP
Feelings about side effects | 1 month after the start of antidepressants treatment
  Patients' feelings about side effects of antidepressants are measured by the FSE
Feelings about side effects | 3 months after the start of antidepressants treatment
  Patients' feelings about side effects of antidepressants are measured by the FSE
Feelings about side effects | 6 months after the start of antidepressants treatment
  Patients' feelings about side effects of antidepressants are measured by the FSE
Satisfaction with treatment | 1 month after the start of antidepressants treatment
  Patients' satisfaction with antidepressants treatment is measured by the SWT
Satisfaction with treatment | 3 months after the start of antidepressants treatment
  Patients' satisfaction with antidepressants treatment is measured by the SWT
Satisfaction with treatment | 6 months after the start of antidepressants treatment
  Patients' satisfaction with antidepressants treatment is measured by the SWT
Satisfaction with information regarding treatment | At the start of antidepressants treatment
  Patients' satisfaction with the received information regarding antidepressants treatment was measured by a sub-scale of the PS-CaTE
Satisfaction with information regarding treatment | 1 month after the start of antidepressants treatment
  Patients' satisfaction with the received information regarding antidepressants treatment was measured by a sub-scale of the PS-CaTE
Satisfaction with information regarding treatment | 3 months after the start of antidepressants treatment
  Patients' satisfaction with the received information regarding antidepressants treatment was measured by a sub-scale of the PS-CaTE
Satisfaction with information regarding treatment | 6 months after the start of antidepressants treatment
  Patients' satisfaction with the received information regarding antidepressants treatment was measured by a sub-scale of the PS-CaTE
Satisfaction with information regarding side effects | At the start of antidepressants treatment
  Patients' satisfaction with the received information regarding side effects of antidepressants was measured by a sub-scale of the PS-CaTE
Satisfaction with information regarding side effects | 1 month after the start of antidepressants treatment
  Patients' satisfaction with the received information regarding side effects of antidepressants was measured by a sub-scale of the PS-CaTE
Satisfaction with information regarding side effects | 3 months after the start of antidepressants treatment
  Patients' satisfaction with the received information regarding side effects of antidepressants was measured by a sub-scale of the PS-CaTE
Satisfaction with information regarding side effects | 6 months after the start of antidepressants treatment
  Patients' satisfaction with the received information regarding side effects of antidepressants was measured by a sub-scale of the PS-CaTE
Health-related quality of life | At the start of antidepressants treatment
  Patients' health-related quality of life is measured by the EQ visual analogue scale from the EQ-5D
Health-related quality of life | 1 month after the start of antidepressants treatment
  Patients' health-related quality of life is measured by the EQ visual analogue scale from the EQ-5D
Health-related quality of life | 3 months after the start of antidepressants treatment
  Patients' health-related quality of life is measured by the EQ visual analogue scale from the EQ-5D
Health-related quality of life | 6 months after the start of antidepressants treatment
  Patients' health-related quality of life is measured by the EQ visual analogue scale from the EQ-5D
Enjoyment and satisfaction | At the start of antidepressants treatment
  Patients' enjoyment and satisfaction is measured by the short-form of the Q-LES-Q
Enjoyment and satisfaction | 1 month after the start of antidepressants treatment
  Patients' enjoyment and satisfaction is measured by the short-form of the Q-LES-Q
Enjoyment and satisfaction | 3 months after the start of antidepressants treatment
  Patients' enjoyment and satisfaction is measured by the short-form of the Q-LES-Q
Enjoyment and satisfaction | 6 months after the start of antidepressants treatment
  Patients' enjoyment and satisfaction is measured by the short-form of the Q-LES-Q

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Liekens, M Psy, Principal Investigator — KU Leuven
Locations (1):
- KU Leuven, Leuven, Vlaams Brabant, Belgium